CLINICAL TRIAL: NCT05098288
Title: Clinical Effectiveness of the MultiCentre Pain Monitor to Guide and Personalize Psychological Treatments: A Single Case Design
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROMEMIUJI
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Emotional Disorder
Keywords: Multicentre Pain Monitor; Transdiagnostic approach; Emotional Disorder; Unified Protocol; Clinical effectiveness

STUDY DESIGN:
Intervention Model Description: Single Case Design (n=1) (multiple baselines)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App + Unified Protocol Arm (Experimental): Participants at this condition will be daily monitored by the app (Multicentre Pain Monitor) while they are administered a self-applied online transdiagnostic intervention (Unified protocol) for their emotional disorders. Alarms will be generated in the face of certain pre-set undesired events.
  Therapists will receive pre-set clinical alarms in real time in the presence of relevant clinical events previously determined by the clinical staff (e.g., clinical worsening or no improvement of functionality, mood or psychological mechanisms worked in therapy). This information will be used to make clinical decisions in a short period of time (e.g., call the patient, or send additional therapeutic material by mail or through the app (momentary ecological intervention), or for its implementation during the course of psychological therapy in order to make the therapy more efficient, safe, personalized and adapted to the needs of the patient
  Interventions: Behavioral: Multicentre Pain Monitor + Unified Protocol

INTERVENTIONS:
Behavioral: Multicentre Pain Monitor + Unified Protocol — The intervention will consist in a self-applied online transdiagnostic intervention for emotional problems together with an app-based EMA. In terms of monitoring, the Multicentre Pain Monitor is a mobile app whose contents have been adapted to conduct ecological momentary assessments in different health conditions. The app assesses important psychological variables, namely anxiety, depressive symptoms,etc. Participants respond daily to the questions in the app. In terms of the online self-applied intervention, the Unified Protocol is a transdiagnostic extension of CBT which works on regulate emotions in a more adaptive way through 5 core treatment modules: present-focused emotional awareness, cognitive flexibility, identification and prevention of emotional avoidance patterns, increasing awareness and tolerance to emotion-elicited physical sensations, and graded (interoceptive and situational) exposure procedures.
  Other Names: Multicentre Pain Monitor

SUMMARY:
The present project aims at testing the clinical effectiveness of an app-based system called Multicentre Pain Monitor for routine outcome monitoring of adult patients with emotional disorders while they are administered a self-applied transdiagnostic psychological intervention (Unified Protocol).

DETAILED DESCRIPTION:
Anxiety and depressive disorders, commonly known as emotional disorders (EDs), are the most frequent mental health problems why patients seek for medical care globally. According to recent epidemiologic studies, lifetime prevalence rates reveal that anxiety and depression disorders affect approximately an estimated 31.9% and 33.7% of people worldwide, respectively. In Spain, a nationwide study showed a prevalence of anxiety and depression disorders of 5.2% and 4.1%, approximately. Consequently, EDs lead to considerable direct and indirect economic losses for countries, as well as a great negative impact on the quality of life and overall functioning of individuals. Adding up to the previous, the current covid-19 pandemic not only has boosted the incidence of mental disorders in healthy people, but also has exacerbated emotional problems in vulnerable populations.

Encouragingly, the effectiveness of psychotherapy for the treatment of EDs, especially cognitive behavioural therapy (CBT), has been supported by a vast amount of scientific evidence. In particular, Internet-delivered CBT (iCBT), where patients sign in to a safe website to access online psychotherapeutic materials within several modules, has emerged in recent years as an effective alternative to face-to-face psychotherapy in an attempt to reduce costs, save therapists' and clients' time, bring psychological treatments closer to the population, and disseminate interventions easily. The growth of digital care has become even more obvious during the covid-19 pandemic and the associated quarantine, where great efforts have been made to adapt evidence-based treatments to a new digital format. Therefore, the current situation has become an opportunity to develop and implement promising digital interventions, which are now more sensible than ever.

To make evidence-based treatments even more accessible, extensions and innovations of CBT have been developed in recent years. The latest research supports a transdiagnostic perspective for the treatment of EDs, where cognitive-behavioural techniques are included to target different EDs altogether. Indeed, the transdiagnostic approach appears to be an effective alternative to single disorder interventions in order to address the high comorbidity rates between anxiety and depressive disorders, as well as the shared mechanisms and the overlapping symptomatology across different disorders which play an essential role in the onset and maintenance of them. In particular, the Unified Protocol (UP), a transdiagnostic extension of CBT which works on regulate emotions in a more adaptive way through different core treatment modules, has been developed for the treatment of EDs. Specifically, the UP shows promising effects not only when delivered onsite, but also online, which makes it an excellent psychological approach to reach a large number of individuals with a single treatment protocol.

In this line, some interesting proposals emphasize the need for a paradigm shift from randomized controlled trials that work on average towards personalized treatments that allow to focus more on the individual (to avoid what group average can mask). In particular, measurement-based care, which consists of routine patient monitoring, periodic feedback to the therapist (or both therapist and patient), and adaptation of the intervention according to such feedback appears to be a feasible option in order to adapt treatments to patients' needs. Fortunately, with the rapid growth of new technologies in our society such as mobile applications (apps), measurement-based care can be implemented more effectively as the apps can be used as support tools for the assessment of several psychological outcome variables. This procedure is commonly known as Ecological Momentary Assessment (EMA) and can help overcome some of the obstacles that traditional, retrospective face-to-face assessments hold. EMA has the potential to assess patients repeatedly and frequently over time, allows to observe fluctuations in patient outcomes, and early interventions can be administered in response to pre-set clinical alarms.

To our knowledge, studies that use technology to improve the management of emotional problems have generally opted for using apps that report on the evolution of treatment to obtain more reliable measures of the evolution of patients or, more frequently, have used different technologies such as web pages or apps to facilitate self-applied treatments based on pre-established modules. The present study goes one step further and explores not only the usefulness of the EMA by means of an app for the improvement of the assessment process of patients with emotional problems/EDs, but also the feasibility of using it to make adjustments in real time or very short-term (e.g., in weekly visits) during the psychotherapeutic process, resembling an ecological momentary intervention (EMI). Several studies have supported the use of EMA to deliver the most personalized feedback or psychological support in real life for a given patient in order to enhance psychotherapy effectiveness and facilitate tailored treatments.

Objectives The current study aims at testing the clinical effectiveness of an app-based system called Multicentric Pain Monitor, which has been recently validated in an empirical study, that monitors individuals with EDs daily and is used as an adjunct tool to the self-applied Internet-delivered transdiagnostic program (UP). The main goal is to explore whether the treatment with the innovative information and communication technologies (ICT) support is effective for persons with emotional disorders.

ELIGIBILITY:
Inclusion Criteria:

* Anxiety or depression problems are the main problematic symptoms
* The patient is over 18 years of age
* The patient is fluent in the language in which the therapy is performed (Spanish in the present study)
* The patient is able to attend to the evaluation and treatment sessions
* The patient signs the informed consent form

Exclusion Criteria:

* The patient presents a severe mental disorder (bipolar disorder, schizophrenia, or an organic mental disorder) or there is suicide risk at the time of assessment
* The patient has used substances in the last three months (excluding cannabis, coffee, and / or nicotine)
* The patient has previously received 8 or more sessions of psychological treatment with clear and identifiable CBT principles in the past 12 months or is currently receiving psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety | Change from baseline to posttreatment. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 0 (not at all) to 3 (completely), "how was your level of anxiety today?"
Change in Depression | Change from baseline to posttreatment. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 0 (not at all) to 3 (completely), "how was your level of depression today?"

SECONDARY OUTCOMES:
Change in Activity level | Change from baseline to posttreatment. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 0 (minimum) to 100 (maximum), "what was your activity level today?"
Change in Emotion Conceptualization | Change from baseline to posttreatment. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 1 (not at all) to 5 (completely), "I see difficult emotions as something bad"
Change in Emotional Avoidance | Change from baseline to posttreatment. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 1 (not at all) to 5 (completely), "Today, I tried to get rid of my unpleasant emotions at all costs"
Change in present-focused emotional awareness (Mindfulness) | Change from baseline to posttreatment. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 1 (not at all) to 5 (completely), "Today, it was easy for me to pay attention to the present moment non-judgmentally"
Change in Cognitive Flexibility | Change from baseline to posttreatment. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 1 (not at all) to 5 (completely), "Today, I was able to consider different interpretations for the bad things that happened to me"
Change in Exposure to situations | Change from baseline to posttreatment. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 1 (not at all) to 5 (completely), "Today, I tried to avoid potentially uncomfortable situations"
Change in Exposure to physical sensations | Change from baseline to posttreatment. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 1 (not at all) to 5 (completely), "Today, I tried to get rid of my unpleasant physical sensations at all costs"

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Gual- Montolio, Study Chair — Universitat Jaume I; Juana Maria Bretón-López, Ph.D., Study Chair — Universitat Jaume I

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with other researchers.